CLINICAL TRIAL: NCT06874023
Title: Warm Up and Cool Down Study: Various Combined Active and Passive Isothermic Heating Protocols, Followed by Different Cooling Protocols, to Increase and Lower Body Core Temperature.
Brief Title: Study to Warm Up and Cool Down Recreationally Active Males Using Different Protocols.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Floris Wardenaar, Assistant Professor, Arizona State University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY00015072
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Heat Acclimation and Thermotolerance
Keywords: Heat; Adaptation; Passive heating

STUDY DESIGN:
Intervention Model Description: Participants performed 4 arms in non-random order (i.e. passive heating, exercise in the heat + passive heating, exercise in the heat, exercise at room temperature), followed by randomized cooling interventions (i.e. a cool slush and one of the three cooling treatments: 1) cool vest, 2) lower arm cool water immersion with cold towel in the neck, 3) combination of 1+2) or heaving no cooling intervention at room temperature with thermoneutral water only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy young men exposed to heating and cooling protocols (Other): All participants underwent four times a heating protocol separated by at least one week, and during these days after undergoing the heating protocol they also participated in a protocol aiming to cool down their body temperature. Each of the four heating and cooling interventions are described as interventions.
  Interventions: Other: Passive heating in hot conditions; Other: Active heating + passive heating in hot conditions; Other: Active heating in hot conditions; Other: Active heating at room temperature; Other: Cool vest; Other: Damp neck towel combined with arm cool water immersion; Other: Combination of cooling interventions; Other: Control in thermoneutral room without cooling

INTERVENTIONS:
Other: Passive heating in hot conditions — Participants performed seated passive heating in 54C conditions
Other: Active heating + passive heating in hot conditions — Participants performed 30 minutes of biking exercise in 43C + 30 min of passive seated heating in 54C conditions.
Other: Active heating in hot conditions — Participants performed 60 minutes of biking exercise in 43C.
Other: Active heating at room temperature — Participants performed active heating through biking exercise for 60 minutes at room temperature.
Other: Cool vest — Cool vest (18°C) with 500 mL (16 fl oz) ice water consumption
Other: Damp neck towel combined with arm cool water immersion — Damp neck towel (24°C) combined with arm (i.e. hand, forearm and half of upper arm) cool water immersion (15°C) and 500 mL (16 fl oz) ice water consumption
Other: Combination of cooling interventions — Combination of cool vest (18°C), damp neck towel (24°C) with arm cool water immersion (15°C), and 500 mL (16 fl oz) ice water consumption
Other: Control in thermoneutral room without cooling — A control with participant sitting in a thermoneutral room (20°C air temperature) without any additional cooling intervention.

SUMMARY:
The objective of this study was to examine the impact of four single-bout heating and cooling strategies on warming up and cooling down core body temperature. Heating strategies included: Passive heating in a hot environment (60 min), Active heating (30 min) + passive heating (30 min) in a hot environment, Active heating(60 min) in a hot environment, and Active heating (60 min) at room temperature. Cooling strategies to reduce body core temperature to baseline included: Cool vest (18°C) , Damp neck towel (24°C) combined with arm (i.e. hand, forearm and half of upper arm) cool water immersion (15°C), Combination of both, A control with participant sitting in a thermoneutral room (20°C air temperature) without any additional cooling intervention.

DETAILED DESCRIPTION:
This semi-randomized crossover control trial was performed between September and October 2020. Data collection took place over the course of 5-weeks with 10 subjects, with one data collection session with all subjects per week (hence, 40 trials total). Baseline gastrointestinal temperature (Tgi) was recorded, and the final Tgi at the end of the heating intervention (Part I), was used as the starting temperature for the current study (Part II).

Part I focused on assessing the efficacy of different heating strategies (Passive heating in a hot environment (60 min), Active heating (30 min) + passive heating (30 min) in a hot environment, Active heating(60 min) in a hot environment, and Active heating (60 min) at room temperature), aiming to reach a core temperature of 38.5°C during a 60-minute period.

Part II focused on cooling the body to a pre-exercise baseline core temperature. Cooling strategies consisted of: 1) Cool vest (18°C) with 500 mL (16 fl oz) ice water consumption, 2) Damp neck towel (24°C) combined with arm (i.e. hand, forearm and half of upper arm) cool water immersion (15°C) and 500 mL (16 fl oz) ice water consumption 3) Combination of cool vest (18°C), damp neck towel (24°C) with arm cool water immersion (15°C), and 500 mL (16 fl oz) ice water consumption or 4) A control with participant sitting in a thermoneutral room (20°C air temperature) without any additional cooling intervention. Thermoneutral water was consumed ad libitum for all interventions in addition to the 500 mL (16 fl oz) ice water consumption for experimental trials (#1-3).

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy
* non-smoking
* uninjured
* active (training five to ten hours per week)

Exclusion Criteria:

* Participants were screened for fitness using the Physical Activity Readiness Questionnaire (PAR-Q): scoring one or more items as a yes.
* Contraindications to use a body core temperature sensor capsule.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Body core temperature | During 60 minute of heating intervention, followed by 60 minutes of cooling intervention.
  A portable telemetry system (E-Celsius, BodyCAP, Hérouville Saint-Clair, France) for temperature sensor capsule, with an accuracy of +/- 0.2°C, was used to measure body core temperature.

SECONDARY OUTCOMES:
Skin temperature | During 60 minute of heating intervention, followed by 60 minutes of cooling intervention.
  Wireless temperature sensors (iButton DS1+2L, Dallas Semiconductor Corp, USA), with an accuracy of ± 0.5°C and a resolution of 0.0625°C, were used to measure Tsk at 20-second intervals. Sensors at four locations (neck, right shoulder, and right shin with all 0.28 weighted coefficient, and left hand with a coefficient of 0.16 to calculate weighted Tsk outcome) as suggested per ISO protocol, held in place at the skin using Opsite transparent film (Opsite Flexigrid, Smith & Nephew Medical Limited, Hull, England).
Heart rate | During 60 minute of heating intervention, followed by 60 minutes of cooling intervention.
  Participants wore an elastic chest strap device (Bioharness-3, Zephyr Technology, Annapolis, MD, USA), measuring HR in beats per minute (bpm) at 1-second intervals.

OTHER OUTCOMES:
Sweat rate | Covering the 60 min of heating and 60 min of cooling resulting in an average sweat rate per hour.
  To determine sweat rate fluid intake, body mass, and urine volume was collected and sweat rate was calculated.
Urine specific gravity | Pre (within 30 min before heating) and post heating (within 5 min after finishing heating) and cooling interventions (within 5 min after finishing cooling).
  As a marker for urine concentration urine specific gravity (USG) was measured.
Environmental temperature | Continuous measurements during the 60 minute heating intervention, followed by the total duration of cooling to baseline intervention for a maximum of 60 minutes.
  During each intervention, the ambient temperature of each testing condition were logged every minute (Kestrel 5400 Heat Stress Tracker with wind vane, Nielsen-Kellerman, Boothwyn, PA, USA).
Relative humidity | Continuous measurements during the 60 minute heating intervention, followed by the total duration of cooling to baseline intervention for a maximum of 60 minutes.
  During each intervention, the relative humidity of each testing condition were logged every minute (Kestrel 5400 Heat Stress Tracker with wind vane, Nielsen-Kellerman, Boothwyn, PA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Community Services Building, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No